CLINICAL TRIAL: NCT02062099
Title: PET Imaging of the Translocator Proteine Ligands (TSPO) With [18 F] DPA-714 Biomarker of NeuroInflammation in Cognitive Decline (NIDECO)
Acronym: NIDeCo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHAO13-CH/ NIDeCo
Record Dates: First submitted 2014-01-17; First posted 2014-02-13 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2014-02

CONDITIONS: Memory Complaint; Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Memory complaint /MCI/ mild to moderate MA (Experimental): Memory complaint (without cognitive decline): 12 patients/ Mild Cognitive Impairment: 12 patients/ Mild to moderate Alzheimer Disease: 12 patients
  Interventions: Drug: [18F]DPA-714 PET/ [18F]AV-45 PET/neuropsychological assessment

INTERVENTIONS:
Drug: [18F]DPA-714 PET/ [18F]AV-45 PET/neuropsychological assessment

SUMMARY:
Alzheimer's disease (AD) is the most common cause of dementia in elderly subjects. AD is characterized by brain lesions like extracellular deposits of ß-amyloïd proteins in senile plaques and intracellular neurofibrillary tangles of hyper-phosphorylated tau protein, both of which are associated with the loss of neurons. The development of disease biomarkers for AD (Tau, PhTau and βamyloid dosing in the cerebrospinal fluid, brain MRI, amyloid PET imaging and fluorodeoxyglucose PET imaging) to identify the pathophysiological processes underlying cognitive impairment biomarkers, have been incorporated into revised diagnosis guidelines.

Post-mortem human AD and AD animal model studies have reported inflammatory processes also implicated in the neuropathology of AD, and upregulated levels of pro-inflammatory cytokines.

In vivo visualization of microglial activation has become possible with the development of molecular imaging ligands (tracers) for use with positron emission tomography (PET). The translocator protein (TSPO) formerly known as the peripheral benzodiazepine receptor (PBR), a receptor located in the outer membrane of mitochondria, is upregulated during neuroinflammation. So targeting TSPO with radiolabeled ligands for PET is considered as an attractive biomarker for neuroinflammation.

The main aim of this pilot study is to quantify neuroinflammation, in terms of fixation and distribution of [18F] DPA-714(Binding Potential BP), and to study its relationship with amyloid load, measured with in [18F]AV-45 (Standard Uptake Values ratio) in cognitive decline.

DETAILED DESCRIPTION:
Molecular imaging of microglial activation could help us document the central inflammatory status of study subjects and assist us in designing future research studies particularly with respect to which subjects to enrol into clinical trials and to evaluate the benefit of specific therapies in selected groups, for example, by monitoring the effects of Aß immunization.

ELIGIBILITY:
Inclusion Criteria:

Criteria common to all participants:

* Signed informed consent
* Age ≥ 60 years old (60-80 years old)
* Native language: French
* Correct sensory abilities (hearing aids accepted) to perform the tests
* Affiliated to a social security system

Criteria for patients with mild to moderate Alzheimer disease defined according to the NINCDS-ADRDA {McKhann, 2011 # 408}:

* MMS between 20 and 25
* contraindication for MRI

Criteria for amnestic MCI patients:

* Amnestic mildcognitive disorder evoking a MA in pre stage dementia {Dubois, 2010 # 273, Dubois, 2007 # 42; Pertersen, 1999 # 21, Albert, 2011 # 409} older than 60 years.

Criteria for patients with isolated memory Complaint (Without Cognitive Decline):

* MMS score ≥ 26
* Normal performance by age and educational level

No inclusion criteria :

* medical history of evolutive disease with conséquences on NCS, chronic alcohol intake, severe depression with MADRS stage > 18
* MA subjects : antagonistic treatment with N-methyl-D-aspartate
* MA or MCI subjects : anomaly on neurologic clinical examination different of the usual symptomatology

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01; Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Fixation and distribution of [18F]DPA-714 (Binding Potential BP) | 2 years
[18F]AV-45 Standard Uptake Values ratio | 2 years

SECONDARY OUTCOMES:
Relationship between [18F]DPA-714 uptake and cognitive, affective symptoms at baseline. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Emilie BEAUFILS, PhD, Principal Investigator — University Hospital of Tours (CMRR)
Locations (1):
- University Hospital of Tours, Tours, France

REFERENCES:
- [Result] Arlicot N, Vercouillie J, Ribeiro MJ, Tauber C, Venel Y, Baulieu JL, Maia S, Corcia P, Stabin MG, Reynolds A, Kassiou M, Guilloteau D. Initial evaluation in healthy humans of [18F]DPA-714, a potential PET biomarker for neuroinflammation. Nucl Med Biol. 2012 May;39(4):570-8. doi: 10.1016/j.nucmedbio.2011.10.012. Epub 2011 Dec 14. PMID 22172392
- [Result] Camus V, Payoux P, Barre L, Desgranges B, Voisin T, Tauber C, La Joie R, Tafani M, Hommet C, Chetelat G, Mondon K, de La Sayette V, Cottier JP, Beaufils E, Ribeiro MJ, Gissot V, Vierron E, Vercouillie J, Vellas B, Eustache F, Guilloteau D. Using PET with 18F-AV-45 (florbetapir) to quantify brain amyloid load in a clinical environment. Eur J Nucl Med Mol Imaging. 2012 Apr;39(4):621-31. doi: 10.1007/s00259-011-2021-8. Epub 2012 Jan 18. PMID 22252372
- [Result] La Joie R, Perrotin A, Barre L, Hommet C, Mezenge F, Ibazizene M, Camus V, Abbas A, Landeau B, Guilloteau D, de La Sayette V, Eustache F, Desgranges B, Chetelat G. Region-specific hierarchy between atrophy, hypometabolism, and beta-amyloid (Abeta) load in Alzheimer's disease dementia. J Neurosci. 2012 Nov 14;32(46):16265-73. doi: 10.1523/JNEUROSCI.2170-12.2012. PMID 23152610
- [Result] Beaufils E, Dufour-Rainfray D, Hommet C, Brault F, Cottier JP, Ribeiro MJ, Mondon K, Guilloteau D. Confirmation of the amyloidogenic process in posterior cortical atrophy: value of the Abeta42/Abeta40 ratio. J Alzheimers Dis. 2013;33(3):775-80. doi: 10.3233/JAD-2012-121267. PMID 22986776
- [Result] Corcia P, Tauber C, Vercoullie J, Arlicot N, Prunier C, Praline J, Nicolas G, Venel Y, Hommet C, Baulieu JL, Cottier JP, Roussel C, Kassiou M, Guilloteau D, Ribeiro MJ. Molecular imaging of microglial activation in amyotrophic lateral sclerosis. PLoS One. 2012;7(12):e52941. doi: 10.1371/journal.pone.0052941. Epub 2012 Dec 31. PMID 23300829